CLINICAL TRIAL: NCT01670812
Title: Clinical Study of Chemoimmunotherapy With Fresh Frozen Plasma, High Dose Methylprednisolone and Rituximab for Ultra-high Risk Chronic Lymphocytic Leukemia
Brief Title: Trial of FFP+HDMP+Rituximab for Ultra-high Risk Chronic Lymphocytic Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-CLL-001
Record Dates: First submitted 2012-08-19; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; ultra-high risk; fresh frozen plasma; methylprednisolone; rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Methylprednisolone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FFP+HDMP+Rituximab (Experimental): Fresh frozen plasma 400ml IV day0, Rituximab: 375 mg/m2 IV day0(after infusion of FFP), methylprednisolone 1g/m2(up to 1.5g) IV day1-day5.
  Interventions: Drug: FFP+HDMP+Rituximab

INTERVENTIONS:
Drug: FFP+HDMP+Rituximab — This is a single arm, multicenter clinical trial, and the regimen including Fresh frozen plasma 400ml IV day0, Rituximab: 375 mg/m2 IV day0(after infusion of FFP), methylprednisolone 1g/m2(up to 1.5g) IV day1-day5
  Other Names: fresh frozen plasma; methylprednisolone; rituximab

SUMMARY:
The purpose of this study is to investigate efficacy and safety of fresh frozen plasma(FFP), high dose methylprednisolone(HDMP) and rituximab for ultra-high risk chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia remains incurable and particularly in ultra-high risk subgroup, and the prognosis of these patients is still dismal.

This is a phase III, multicenter perspective clinical trial of combination of fresh frozen plasma(FFP), high dose methylprednisolone(HDMP) and rituximab for ultra-high risk chronic lymphocytic leukemiaThe. The main purpose of this study is to investigate efficacy and safety of this combinated regimen in subgroup of CLL patients.

All the enrolled patients will be followed during and after the treatment period up to one year. Interim and final evaluation will be done after each cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years old.
2. Diagnosis of chronic lymphocytic leukemia.
3. Active disease meeting at least one of the International Workshop on Chronic Lymphocytic Leukemia 2008 criteria for requiring treatment.
4. Ultra-high risk CLL(Meets at least one of the following criteria) (1)ultra high-risk genetics (17p deletion and/or TP53 mutation) (2)short PFS(<24 months)after intense immunochemotherapy treatment(i.e. FCR, FR, PCR, BR etc) (3)fludarabine-refractory
5. Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Severe allergic constitution or asthma.
2. Recent myocardial infarction or hypotension.
3. ECOG performance status of ≤ 2 at study entry.
4. Active hepatitis B(DNA >1×103/ml)
5. Severe and uncontrolled diabetes mellitus.
6. Severe and uncontrolled hypertension(BP> 150/90 mmHg after treatment).
7. Active and uncontrolled systematic infection which need treatment of antibiotics.
8. Clinical symptoms of dysfunction of central nervous system.
9. Unstable and severe gastrorrhagia and peptic ulcer.
10. Major surgery within three weeks.
11. Any potential drug abuse, medical, psychological or social conditions which may disturb this investigation and assessment.
12. In any conditions which investigator considered ineligible for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
overall response rate | one year
  overall response rate after treated by FFP+HDMP+Rituximab regimen

SECONDARY OUTCOMES:
progression free survival | one year
  progression free survival after treatment of FFP+HDMP+Rituximab for ultra-high risk CLL patients.
overall survival | one year
  overall survival after treatment of FFP+HDMP+Rituximab for ultra-high risk CLL patients
Number of Participants with Adverse Events | up to 30 days after last dose of treatment
  Number of Participants with Adverse Events, and evaluated standard is according to common terminology criteria adverse events(CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (14):
- China (14):
  - The First affiliated Hospital of AnHui Medical Universtiy, Hefei, Anhui
  - TongJi Hospital, Wuhan, Hubei
  - ChangZhou First People's Hospital, Changzhou, Jiangsu
  - ChangZhou No.2 People's Hospital, Changzhou, Jiangsu
  - HuaiAn First People's Hospital, HuaiAn, Jiangsu
  - NanJing First People's Hospital, Nanjing, Jiangsu
  - JiangSu Province Hospital, Nanjing, Jiangsu
  - JiangSu Province Hospital of TCM, Nanjing, Jiangsu
  - WuXi People's Hospital, Wuxi, Jiangsu
  - ZhenJiang First People's Hospital, Zhenjiang, Jiangsu
  - Shandong Provincial Hospital, Jinan, Shandong
  - TongJi Medical University affiliated TongJi Hospital, Shanghai, Shanghai Municipality
  - West China School of Medicine, West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Background] Xu W, Miao KR, Zhu DX, Fang C, Zhu HY, Dong HJ, Wang DM, Wu YJ, Qiao C, Li JY. Enhancing the action of rituximab by adding fresh frozen plasma for the treatment of fludarabine refractory chronic lymphocytic leukemia. Int J Cancer. 2011 May 1;128(9):2192-201. doi: 10.1002/ijc.25560. PMID 20635386
- [Background] Xu W, Miao KR, Hong M, Zhu DX, Fang C, Dong HJ, Wang DM, Cao X, Li JY. High-dose methylprednisolone can induce remissions in patients with fludarabine-refractory chronic lymphocytic leukaemia. Eur J Cancer. 2010 Aug;46(12):2145-9. doi: 10.1016/j.ejca.2010.04.021. Epub 2010 Jun 4. PMID 20627536
- [Background] Dungarwalla M, Evans SO, Riley U, Catovsky D, Dearden CE, Matutes E. High dose methylprednisolone and rituximab is an effective therapy in advanced refractory chronic lymphocytic leukemia resistant to fludarabine therapy. Haematologica. 2008 Mar;93(3):475-6. doi: 10.3324/haematol.11903. PMID 18310545
- [Background] Klepfish A, Gilles L, Ioannis K, Rachmilewitz EA, Schattner A. Enhancing the action of rituximab in chronic lymphocytic leukemia by adding fresh frozen plasma: complement/rituximab interactions & clinical results in refractory CLL. Ann N Y Acad Sci. 2009 Sep;1173:865-73. doi: 10.1111/j.1749-6632.2009.04803.x. PMID 19758239